CLINICAL TRIAL: NCT06392555
Title: Fetal Heart Ultrasound Suspicious Radiographic Finding Identification - Reader Study
Status: Completed | Type: Observational
Sponsor: BrightHeart (Industry)
Responsible Party: Sponsor
Other Study IDs: reader2024
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Prenatal ultrasound examinations
  Interventions: Device: Device-Aided performances; Other: Device-Unaided performances

INTERVENTIONS:
Device: Device-Aided performances — Determination of the presence of the 8 findings suspicious of CHD by readers, aided by the device
Other: Device-Unaided performances — Determination of the presence of the 8 findings suspicious of CHD by readers, unaided by the device

SUMMARY:
Clinical performance of the device will be evaluated in a fully-crossed, multiple-reader multiple-case (MRMC) study. This study will be used to determine the impact of the device on reader performance in identifying suspicious radiographic findings in fetal heart ultrasound video clips recorded during 2nd trimester anatomic ultrasound examinations conducted during the second trimester of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* ultrasound examinations conducted during the second trimester of the pregnancy
* fetus between 18 and 24 weeks of gestational age
* mothers 18 years old or older

Exclusion Criteria:

* exams corresponding to multiple pregnancy
* fetal heterotaxy
* exams not containing video clips with interpretable 4-chamber (4C), Left Ventricular Outflow Tract (LVOT) or Right Ventricular Outflow Tract (RVOT) standard views

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ultrasound examinations conducted during the second trimester of the pregnancy, containing interpretable 4-chamber, LVOT and ROVT standard views of the fetal heart
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
AUC of the ROC curve for the presence of any suspicious finding | 1 month
  AUC of the ROC curve for both reading conditions (aided vs unaided by the device) derived from the identification of any suspicious radiographic finding

SECONDARY OUTCOMES:
AUC of the ROC curve for the presence of each suspicious finding | 1 month
  AUCs of the ROC curve for both reading conditions (aided vs unaided by the device) for identification of each finding.
Sensitivity and specificity for both reading conditions for the presence of any suspicious finding | 1 month
  Sensitivity and specificity for both reading conditions (aided vs unaided by the device) for identification of each finding.
Sensitivity and specificity for both reading conditions for the presence of each suspicious finding | 1 month
  Sensitivity and specificity for both reading conditions for the presence of each suspicious finding.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Gardella, PhD, Study Director — Chief Technical Officer
Locations (1):
- MFM Associates, PLLC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
no sharing of the IPD is planned